CLINICAL TRIAL: NCT00736112
Title: A New Approach to Otitis Media With Effusion (OME)
Brief Title: Food Allergy - Tubes - Adenoids (FATA) Trial
Acronym: FATA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator left the institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-ENT- 1120277
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Otitis Media With Effusion; Food Hypersensitivity
Keywords: Food Allergy in Children; Otitis Media with Effusion (OME); Recurrent Middle Ear Infections; Middle Ear Fluid; Food Allergy and Otitis Media with Effusion; Recurrent middle ear fluid in children <4 years old; Chronic ear infections in children <4 years old
MeSH Terms: conditions — Otitis Media with Effusion; Food Hypersensitivity | interventions — Adenoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMT and food allergy (Experimental): trial subjects will receive food allergy testing and management in conjunction with BMT (Bilateral Myringotomy with Tympanostomy Tubes). Food allergy management involves parental education on how to avoid the specific offending foods.
  Interventions: Other: Food Allergy Testing; Procedure: BMT
- BMT and adenoidectomy (Experimental): involves BMT (Bilateral Myringotomy with Tympanostomy Tubes), adenoidectomy, and food allergy testing and management.
  Food allergy management involves parental education on how to avoid the specific offending foods.
  Interventions: Other: Food Allergy Testing; Procedure: Adenoidectomy; Procedure: BMT
- BMT alone (Active Comparator): The standard protocol for children presenting with initial Chronic OME is to perform a BMT (Bilateral Myringotomy with Tympanostomy Tubes).
  Interventions: Procedure: BMT

INTERVENTIONS:
Other: Food Allergy Testing — Food Allergy Diagnosis - blood drawn for food allergy testing at the time of surgery (bilateral myringotomy with tympanostomy tubes +/- adenoidectomy)
  Arms: BMT and adenoidectomy; BMT and food allergy
Procedure: Adenoidectomy — Adenoidectomy to remove adenoid tissue. (Are adenoids a factor in OME (otitis media with effusion) or is food allergy diagnosis and treatment able to significantly prevent ROM (recurrent otitis media) after the tubes fall out?)
  Arms: BMT and adenoidectomy
Procedure: BMT — The standard protocol for children presenting with initial Chronic OME is to perform a BMT
  Other Names: Bilateral myringotomy with tympanostomy tubes

SUMMARY:
The questioned proposed by this study is one of treatment: "To what extent does simultaneous BMT (Bilateral Myringotomy with Tympanostomy Tubes), adenoidectomy, and diagnosis/avoidance of food allergy affect the frequency of recurrent otitis media (ROM) versus the standard academy approach (tube insertions only) to chronic otitis media with effusion; furthermore, are adenoids a factor in OME or is food allergy diagnosis and treatment able to significantly prevent ROM after the tubes fall out?"

The trial seeks to provide evidence that the treatment for Chronic OME in children should involve surgical procedures (BMT +/- adenoidectomy), as well, as a food allergy work-up and subsequent avoidance of the offending foods in order to significantly decrease ROM.

To answer this question, a prospective, randomized controlled trial needs to be conducted. Since a majority of OME patients are from the pediatric population, parental consent must be obtained. Subjects in our study will initially present to the clinic with otitis media symptoms and diagnostic tests such as a tympanogram, otoscopy, and history of recurrent otitis media will be obtained. Once the surgical decision for bilateral myringotomy and tympanostomy tubes has been made, parents will be informed about the trial. The standard protocol for children presenting with initial Chronic OME is to perform a BMT. Therefore, data from the control group (Group 1) will be obtained from faculty ENT who follow the academy's recommendations. Data from Group 2 and 3 will be collected from other ENT faculty members, including the faculty co-investigator who will perform the BMT and obtain a food allergy blood draw at the time of surgery. The study's faculty co-investigator will describe food avoidance techniques to post-op patients from Groups 2 and 3. Patients with previous adenotonsillar surgery or placement of tympanostomy tubes will not be enrolled in the study. The incidence of ROM episodes in all trial groups will be recorded.

DETAILED DESCRIPTION:
Design: Randomized controlled trial to evaluate the efficacy of a new approach in the treatment of children presenting with chronic otitis media with effusion. The new approach calls for a surgical correction of OME by a BMT (Bilateral Myringotomy with Tympanostomy Tubes) +/- Adenoidectomy, with additional food allergy diagnosis and subsequent management of offending foods in order to reduce the frequency of recurrent otitis media (ROM).

End Points: Comparison between groups (1,2,3) on the recurrence of otitis media following surgery. All trial participants will have follow-up clinic appointments every three months until tubes fall out and after this point, patients will present to clinic every three months for one year for evaluation of recurrent middle ear fluid. Questionnaires will be administered to Groups 2 & 3 at the F/U appointments to evaluate food allergy management.

Methodology: Trial participants will be identified by their otitis media signs and symptoms. Subjects who meet the inclusion criteria will be asked to participate in the study and consent will be obtained. Surgery will be performed based on group assignment. All trial subjects will receive standard post-op care and will also be seen for clinical evaluation q 3 months post-surgery, and then q 3 months after the tubes are out for one year. The number of otitis media episodes during the follow up year in children assigned to groups 1,2, and 3 will be recorded.

Procedures: At the initial clinic visit, potential trial subjects will be asked about their otitis media history, including how many episodes of OM in the past six months, evidence of hearing loss, lack of response to antibiotic therapy, prolonged periods of OME, and previous tympanograms. Pediatric patients will have their tympanic membranes (TM) evaluated by otoscopy for evidence of OME. Tympanometry will also be performed to confirm the presence of fluid in the middle ear.

Participants in the control group (Group 1) will receive the standard academy regimen for initial presentation of Chronic OME, which is insertion of BMT. Group 2 trial subjects will receive food allergy testing and management in conjunction with BMT. Group 3 involves BMT insertion, adenoidectomy, and food allergy testing and management.

Food management involves parental education on how to avoid the specific offending foods by their allergic children.

The total length of subject participation is variable depending on when the tubes come out. Once the tubes have fallen out, the patient will be evaluated every three months for one full year.

ELIGIBILITY:
Inclusion Criteria:

1. Otoscopy reveals Chronic OME.
2. Tympanometry confirms fluid in middle ear.
3. Children <4 years old
4. Lack of improvement after three months of antibiotic therapy.
5. History of persistent effusion for three or more months per-episode of OM.
6. >3 episodes of AOM in preceding 6 months or >5 episodes of AOM during preceding 12 months
7. Bilateral conductive hearing loss of 15 dB or more.

Exclusion Criteria:

1. Previous adenotonsillar surgery or placement of tympanostomy tubes.
2. Children with inhalant allergies including asthma.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The number of post-op ROM episodes in each group (1,2,3) will be recorded throughout the study (after the tympanostomy tubes fall out). | Trial participants will have follow-up appointments every three months until tubes fall out, then patients will have F/U every three months for one year for evaluation of recurrent middle ear fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Young Paik, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital: Department of Otolaryngology - Head and Neck Surgery, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No